CLINICAL TRIAL: NCT06809231
Title: Effectiveness and Safety of Knee Cartilage Lesion Treatment Using CartiONE: 1-to-13 Year Follow-up
Acronym: ICONIC
Status: Recruiting | Type: Observational
Sponsor: Cartilage Repair Systems BV (Industry)
Responsible Party: Sponsor
Other Study IDs: CRS001-2023; IRAS ID 345492 (Other: IRAS)
Record Dates: First submitted 2025-01-17; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Knee Cartilage Lesion
Keywords: knee cartilage; CartiONE; ICONIC; coimplantation; chondron; one stage; intraoperative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated with CartiONE

SUMMARY:
CartiONE is a technique used in autologous articular-chondrocyte-based treatments for symptomatic focal articular-cartilage lesions of the knee. The CartiONE technique was evaluated in combination with an osteochondrally placed, biodegradable, biocompatible, load-bearing copolymer (PolyActive) scaffold in the INSTRUCT trial (NCT01041885). To evaluate the clinical effectiveness of the CartiONE technique and confirm its safety, in this study retrospective baseline data and follow-up data, documented as per the standard of care at the participating hospitals, will be collected for patients who were treated with CartiONE.

The potential number of patients in this study is 122 and involves patients treated with CartiONE from 2010 to 2023 with a minimum follow-up period of six months, spread across five countries: Belgium, England, Greece, Poland, and Austria.

DETAILED DESCRIPTION:
Inclusion and exclusion criteria Inclusion criteria Patients treated with CartiONE for knee cartilage lesion more than 6 months prior to inclusion in this study.

The study site holds a patient record of all relevant medical history data, including operation reports of any prior knee surgeries, the index knee surgery report, and posttreatment observations and re-intervention reports, if applicable.

Exclusion criterion Patients cannot be included if any condition exists that is judged by the treating surgeon as making the patient not suited for participation.

Statistics This is a retrospective, open label, non-randomized, single arm trial. Since different questionnaires for effectiveness and for quality of life (e.g., KOOS, EQ-5D,…) may have been used, the total score of the questionnaires ranging from the minimum total score (i.e. 0 or 1) to the maximum total score will be transformed into the range from 0 respective 1 to 100. Now they can be combined across patients and effectiveness questionnaires or across patients and quality of life questionnaires. Details will be provided in the Statistical Analysis Plan.

There are two co-primary endpoints:

Primary endpoint safety:

Adverse events with particular focus on Treatment failure rate and on other AESIs

Primary endpoint effectiveness:

MOCART sub-score 1 "Volume fill of cartilage defect"

Efficacy/Effectiveness:

Key secondary endpoints:

Non-inferiority in MOCART/MOCART 2.0 total scores when measured at two different visits, i.e., at the reference visit and later.

Non-inferiority in mean "Radiologist's overall knee status assessment" when measured on a scale from 0 (extremely bad) to 100 (extremely good) at two different visits, i.e., at the reference visit and later.

Other secondary endpoints:

Improvement in other effectiveness questionnaire total scores Improvement in quality-of-life total scores Improvement in other questionnaires when applicable

Exploratory endpoint:

"Radiologist's overall knee status assessment" on a scale from 0 (extremely bad) to 100 (extremely good) of the two readers.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with CartiONE for knee cartilage lesion more than 6months prior to inclusion in this study.
* The study site holds a patient record of all relevant medical history data, including operation reports of any prior knee surgeries, the index-knee surgery report, and posttreatment observations and re-intervention reports, if applicable.

Exclusion Criteria:

* Patients cannot be included if any condition exists that is judged by the treating surgeon as making the patient not suited for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with CartiONE for knee cartilage lesions
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events with particular focus on Treatment failure rate and on other AESIs | periprocedurally, through to study completion up to 2 years
MOCART sub-score 1 "Volume fill of cartilage defect" | baseline, month 3, month 6, year 1, year 2

CONTACTS AND LOCATIONS:
Locations (5):
- Belgium (2):
  - UZ Ghent, Ghent, Oost-Vlaanderen
  - AZ Monica, Antwerp
- MIRAI, Warsaw, Poland
- United Kingdom (2):
  - University Hospitals Coventry & Warwickshire NHS Trust, Coventry
  - Robert Jones & Agnes Hunt Orthopaedic Hospital NHS Foundation Trust, Oswestry

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://cartione.com/